CLINICAL TRIAL: NCT06763211
Title: Effect of Chlorhexidine Gluconate Hair Bath on the Development of Surgical Site Infection and Time to Discharge in Patients Scheduled for Cranial Surgery: Randomized Controlled Study
Brief Title: Effect of Chlorhexidine Gluconate Hair Bath on the Development of Surgical Site Infection and Time to Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HAVVA ÇOŞKUN (Other)
Collaborators: Serpil İNCE (Unknown)
Responsible Party: Sponsor-Investigator, HAVVA ÇOŞKUN, Akdeniz University, Akdeniz University Hospital
Organization: Akdeniz University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AkdenizNeurology
Record Dates: First submitted 2024-04-29; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Infection Secondary to Surgical Procedure
Keywords: Cranial surgery; Surgical site infection; Hair bath; chlorhexidine gluconate
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled, single-blind experimental study. The sample will be divided into three groups in total, two intervention groups and one control group, by randomization method. The intervention 1 group will have a hair bath with chlorhexidine the evening before the operation, the intervention 2 group will first have a hair bath with the product used by the patient and then with chlorhexidine, and the control group will have a hair bath with the soap/shampoo the patient uses himself. The product available on the market will be used. The hair of patients in intervention groups 1 and 2 will be washed twice, using 5 ml of chlorhexidine each time. After applying the solution, it will be left for 1 minute and then rinsed. After rinsing, the hair will be dried with a disposable towel.
Who Masked: Participant
Masking Description: Statistics Expert
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Experimental): Hair bath will be applied to the patient by the researcher. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. Hair bath will be done with 5 ml chlorhexidine gluconate solution at the patient's bed. After the hair is wetted, chlorhexidine gluconate will be applied to the entire scalp and hair, the scalp and hair will be rubbed with gentle movements for 5 minutes and left for 1 minute before rinsing. Application of the solution will be repeated twice. It will be rinsed after waiting for a minute. It will be dried with disposable towels. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.
  Interventions: Procedure: Chlorhexidine Hair Bath
- Intervention 2 (Experimental): Hair bath will be applied to the patient by the researcher. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. First, the researcher will give a hair bath using the patient's soap or shampoo. In the same way, it will be rubbed for 5 minutes and left for 1 minute before rinsing. Secondly, the patient will be given a hair bath with 5 ml of chlorhexidine gluconate solution. It will be rubbed with chlorhexidine gluconate for 5 minutes and left for 1 minute before rinsing. Application of the solution will be repeated twice. The patient's hair will be dried with a disposable towel. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.
  Interventions: Procedure: Chlorhexidine Hair Bath
- Control (No Intervention): Hair bath will be applied to the patient by the researcher. Hair bath will be given using the patient's own soap or shampoo. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. The soap or shampoo will be applied to the scalp and hair by rubbing with gentle movements for 5 minutes and then left for one minute. After the hair and scalp are rinsed, they will be dried with disposable towels. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.

INTERVENTIONS:
Procedure: Chlorhexidine Hair Bath — Intervention group 1 will have a hair bath with 5 ml of chlorhexidine gluconate solution 2 times consecutively. Intervention group 2 will first be given a hair bath using the patient's soap or shampoo. Afterwards, the hair will be bathed 2 times consecutively with 5 ml chlorhexidine gluconate solution. Hair bath will be given to the control group using the patient's own soap or shampoo. Surgical site infection follow-up form, laboratory findings form, vital signs form, culture follow-up form will be filled out before and after banyadon. Additionally, cultures will be taken from the surgical area with hair immediately after bathing, on the 2nd post-operative day, and on the day the stitches are removed.
  Arms: Intervention 1; Intervention 2

SUMMARY:
One of the most important preventable complications occurring in the postoperative period is surgical site infections. Surgical site infections (SSI) are infections that occur in incisions, organs or organ spaces that occur after surgery. The mortality rate of patients who develop SSI is twice as high as that of patients who do not develop infection, the duration of intensive care stay increases by 60%, and the rate of hospital admission after discharge is five times higher. As the number of surgical procedures and procedures continues to increase, preventing surgical site infections becomes increasingly important. One of the reasons for infection after cranial surgery is the patient's scalp flora. The skin and scalp have the potential to cause many bacterial and harmful fungal infections. The Center for Disease Control and Prevention (CDC) recommends that patients take a shower/bath with soap or an antiseptic solution at least one night before the day of surgery. Although there is no definitive evidence that this practice reduces surgical site infections, the fact that most surgical site infections are caused by microorganisms on the skin supports the recommendation.

The research was planned as a randomized controlled, single-blind experimental study. The sample will be divided into three groups in total, two intervention groups and one control group, by randomization method. The intervention 1 group will have a hair bath with chlorhexidine the evening before the operation, the intervention 2 group will first have a hair bath with the product used by the patient and then with chlorhexidine, and the control group will have a hair bath with the soap/shampoo the patient uses himself. The product available on the market will be used. The hair of patients in intervention groups 1 and 2 will be washed twice, using 5 ml of chlorhexidine each time. After applying the solution, it will be left for 1 minute and then rinsed. After rinsing, the hair will be dried with a disposable towel.

The purpose of this study; The aim of this study is to evaluate the effect of hair bath with chlorhexidine solution on the occurrence of SSI and discharge time in patients scheduled for cranial surgery in the brain and neurosurgery clinic.

DETAILED DESCRIPTION:
This study; It is thought that it will increase the awareness of nurses about preoperative shower/bath and hair bath in brain and neurosurgery clinics, help the implementation of shower/bath and hair bath protocols in clinics, and be effective in preventing surgical site infections.

The research was planned to determine the effect of hair bath using soap/shampoo, chlorhexidine gluconate solution and both in the evening before surgery on surgical site infection and discharge time in preventing surgical site infection on the scalp in patients scheduled for cranial surgery.

UNIQUE VALUE:

This research will be conducted based on the following hypotheses:

H0_1: Chlorhexidine gluconate hair bath has no effect on the development of surgical site infection in patients planned for cranial surgery.

H 1_1: Chlorhexidine gluconate hair bath has an effect on the development of surgical site infection in patients planned for cranial surgery.

H0_2: Chlorhexidine gluconate hair bath has no effect on the time to discharge in patients planned for cranial surgery.

H1_2: Chlorhexidine gluconate hair bath has an effect on the duration of discharge in patients planned for cranial surgery.

The research is a randomized controlled, single-blind experimental research design.

The population of the research will consist of patients scheduled for cranial surgery at Akdeniz University Hospital Brain and Nerve Surgery Clinic. The sample of the study will consist of patients who meet the inclusion criteria for cranial surgery planned at Akdeniz University Hospital Brain and Nerve Surgery Clinic. In order to calculate the sample size, the power of the study, type 1 error, and effect size parameters were determined with the guidance of similar study data. The sample size was calculated with the support of a statistical consultant. G*Power 3.1.9.4 in calculating the sample size. statistical program was used. In this program, a total of 224 individuals were determined, including 75 intervention 1 group, 75 intervention 2 group, and 74 control group, with an effect size of 96%, 80% power and a margin of error of 0.05. Considering the possibility of sample loss in the study with statistical consultancy, 10% more of the calculated sample was included in the randomization process. It was decided to include a total of 252 people in randomization: 84 in the intervention 1 group, 84 in the intervention 2 group, and 84 in the control group.

This study is planned to be conducted with patients admitted to Research Akdeniz University Hospital Brain and Nerve Surgery Clinic for planned cranial surgery. Patients who meet the planned inclusion criteria for cranial surgery will continue to be included in the study until the sample size is reached. The collection of data in the groups and the implementation of nursing interventions will be carried out by the researcher by meeting the patients face to face. After patients scheduled for cranial surgery are admitted to the clinic, information about the research will be given in the patient room, informed consent will be obtained and an implementation plan will be made. For patients scheduled for cranial surgery who agree to participate in the study and meet the inclusion criteria, the Patient Descriptive Characteristics and Preoperative Period Information Form will be filled out by the researcher together with the patient. The Surgical Site Infection Follow-up Form will be filled out daily by the investigator while observing the cranial surgical area. Laboratory Findings Form, Vital Signs Form and Culture Follow-up Form will be written by the researcher by following the nurse observation forms and the computer system where the patient data are recorded. It is planned to give brochures regarding the care of the surgical field to patients and their relatives before discharge. Patients included in the research will be assigned to groups by a simple randomization method by a statistician outside the thesis.

1. Research Application Steps for Patients in Intervention 1 Group: Hair bath will be applied to the patient by the researcher. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. Hair bath will be done with 5 ml chlorhexidine gluconate solution at the patient's bed. After the hair is wetted, chlorhexidine gluconate will be applied to the entire scalp and hair, the scalp and hair will be rubbed with gentle movements for 5 minutes and left for 1 minute before rinsing. Application of the solution will be repeated twice. It will be rinsed after waiting for a minute. It will be dried with disposable towels. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.
2. Research Application Steps for Patients in Intervention 2 Group: Hair bath will be applied to the patient by the researcher. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. First, the researcher will give a hair bath using the patient's soap or shampoo. In the same way, it will be rubbed for 5 minutes and left for 1 minute before rinsing. Secondly, the patient will be given a hair bath with 5 ml of chlorhexidine gluconate solution. It will be rubbed with chlorhexidine gluconate for 5 minutes and left for 1 minute before rinsing. Application of the solution will be repeated twice. The patient's hair will be dried with a disposable towel. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.
3. Research Application Steps for Patients in the Control Group: Hair bath will be applied to the patient by the researcher. Hair bath will be given using the patient's own soap or shampoo. Before the hair bath, the patient's eyes will be covered with gauze and cotton tampons will be used for the ears. The soap or shampoo will be applied to the scalp and hair by rubbing with gentle movements for 5 minutes and then left for one minute. After the hair and scalp are rinsed, they will be dried with disposable towels. A swab of 2 cm2 will be taken from the scalp with a culture stick by rolling it back and forth for 15 seconds. An area of 2 cm2 will be taken from the area where the patient will be surgically cut.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Having elective surgery
* The patient agrees to participate in the study
* Having cranial surgery for the first time
* No irritated open wound on the scalp
* No systemic infection such as sepsis, pneumonia, blood infections or intracranial infection such as meningitis or abscess
* Not having a mental illness that would prevent communication

Exclusion Criteria:

* Be under 18 years of age
* There is deterioration in the integrity of the cranium and emergency cranial surgery is planned
* Not volunteering to participate in the research
* Having received oncological treatment
* Having a systemic or intracranial infection
* Transsphenoidal surgical intervention is planned
* Having a mental illness that prevents communication
* Being allergic to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Culture Tracking Form | First culture taken at preop morning after hair bath, second culture taken on 2nd postop day, and 3rd culture taken just before surgical site stitches removed 12th day
  Within the scope of the research, the date of culture taken from the surgical area will be recorded and will be used to follow up the results. The culture collection times were after washing, on the 2nd post-operative day, and on the 12th day after the stitches were removed. or 15th day]. The last culture sample will be taken on the day the stitches are removed.
Surgical Site Infection Follow-up Form | It will be applied every day (once a day), starting from the 2nd postoperative day to 7th postoperative day.
  This form, created by the researcher using the relevant literature, consists of two parts. In the first section, there are 17 questions that include patients' data regarding the operation and surgical field. Surgery performed, date, time, duration, duration of stay in intensive care, duration of hospital stay after surgery, date of discharge, duration of antibiotic use, steroids, immunosuppressive and antidiabetic drugs used, postoperative blood transfusion, number and type of drains, withdrawal time, culture from the wound site. It includes questions about the date of collection, how the patient was treated for discharge in the surgical area, whether there is infection in the surgical area, culture results, and the presence of repeated hospitalization
Length of hospital stay | Until Primary Completion is completed. up to 15 days
  The patient's hospital stay will be evaluated with data from patient records, covering the period from the first day of hospitalization to when the patient leaves the clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No